CLINICAL TRIAL: NCT01348854
Title: A Multi-Center Prospective Study to Evaluate the Safety and Effectiveness of Arcuate Incisions Performed With the IntraLase iFS Femtosecond Laser System
Brief Title: Safety and Effectiveness of Arcuate Incisions Performed With the iFS Femtosecond Laser System
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott Medical Optics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMTO-103-ISAK
Record Dates: First submitted 2011-05-04; First posted 2011-05-06 (Estimated); Results first posted 2014-06-04 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-05

CONDITIONS: Corneal Astigmatism
Keywords: astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Natural Astigmatism (Experimental): Use of the iFS Femtosecond Laser System to make arcuate incisions to correct naturally occurring corneal astigmatism in eyes with no prior history of ophthalmic surgery. May include eyes with cataracts.
  Interventions: Device: iFS Femtosecond Laser System
- Post Cataract with Residual Astigmatism (Experimental): Use of the iFS Femtosecond Laser System to make arcuate incisions to correct residual astigmatism in eyes that have undergone cataract extraction. May also include eyes with residual astigmatism following implantation of a phakic intraocular lens implanted.
  Interventions: Device: iFS Femtosecond Laser System

INTERVENTIONS:
Device: iFS Femtosecond Laser System — arcuate incisions placed with the iFS femtosecond laser

SUMMARY:
To determine if arcuate incisions performed with the iFS femtosecond laser are safe and effective in reducing corneal astigmatism.

DETAILED DESCRIPTION:
Surgeons will perform arcuate incisions in the cornea in arc segment patterns using the iFS femtosecond laser to treat subjects with corneal astigmatism.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, of any race, and at least 21 years of age at the time of pre-op exam
2. Corneal astigmatism, as determined by topographic keratometry, of 0.75 D to 4.00 diopters (D)
3. Best Spectacle Corrected Distance Visual Acuity (BSCVA)

   1. Group 1:

      * Natural astigmatism, no cataract - BSCVA of 20/25 or better
      * Pre cataract or phakic IOL surgery - no BSCVA criteria
   2. Group 2:

      * Post IOL surgery- BSCVA of 20/25 or better
4. Uncorrected Visual Acuity (UCVA) of 20/40 or worse
5. Demonstration of agreement: Corneal astigmatism (as determined by topographic keratometry) must be in agreement with refractive astigmatism (as determined by manifest refractions) within </= 0.75 D in magnitude and 15 degrees axis when cylinder </= 1.5 D or 10 degrees axis when cylinder > 1.5 D.
6. Preoperative central pachymetry of >/=480 um
7. Keratometry between 38.0 D (flat) to 48.0 D (steep)
8. Corneal power (diopters) difference at the 3mm point from topographic center shall be </= 1D at the steepest meridian
9. Intraocular pressure of 12 to 21 mm Hg with no glaucomatous retinal/optic nerve changes
10. Subjects who have worn a contact lens within the past 30 days must remove the soft lens at least 2 weeks prior and a rigid or toric lens at least 3 weeks prior to baseline measurements
11. Willing and capable of returning for follow-up examinations for the duration of the study

Exclusion Criteria:

1. Angle kappa of greater than 0.5 mm, absolute value
2. Prior implantation of toric or multifocal intraocular lens
3. Women who are pregnant, breast-feeding, or intend to become pregnant over the course of the study
4. Concurrent use of topical or systemic medications that may impair corneal wound healing
5. History of any ocular or medical conditions that could affect corneal wound healing
6. History of active or recurrent ophthalmic disease, including corneal dystrophy or other non-refractive abnormality such as exposure keratitis or clinically significant dry eye
7. Abnormal topography, including evidence of keratoconus or pellucid marginal degeneration in either eye
8. Evidence of clinically significant corneal opacity/scar in the operative eye(s) within an 8 mm diameter zone of the visual axis
9. Known sensitivity or inappropriate responsiveness to any of the medications used in the post-operative course
10. Participation in any other conflicting clinical study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-05; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Tarantino, OD, Study Director — Abbott Medical Optics
Locations (4):
- Paracelsus Medizinische Privat-Universitat, PMU, Salzburg, Salzburg, Austria
- CHU Morvan, Brest, Brest, France
- Germany (2):
  - Bochum-Langendreer, Bochum, Bochum
  - Potsdamer Augenklinik im, Potsdam, Potsdam

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Natural Astigmatism | Post Cataract With Residual Astigmatism
Started | 34 (53 eyes of 34 participants) | 6 (10 eyes of 6 participants)
Completed | 31 (47 eyes of 31 participants) | 5 (9 eyes of 5 participants)
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Data analysis was performed for eyes treated. Subjects may have had one or both eyes treated. If both eyes, one eye may have been in Natural Astigmatism group and the other eye in the Post Cataract with Residual Astigmatism group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Natural Astigmatism | Post Cataract With Residual Astigmatism | Total
Number analyzed (Participants) | 34 | 6 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (16.6) | 55.0 (15.9) | 53.7 (16.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 5 | 31
  Male | 8 | 1 | 9
Region of Enrollment [Number; unit: paticipants]
  France | 0 | 1 | 1
  Austria | 17 | 2 | 19
  Germany | 17 | 3 | 20

OUTCOME MEASURES:

1. Primary Outcome: Reduction of Astigmatism
Description: Reduction of astigmatism as determined by manifest refractive cylinder
Time Frame: 6 months
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: diopter
Units Other Than Participants: eyes
Arm/Group | Natural Astigmatism | Post Cataract With Residual Astigmatism
Number analyzed (Participants) | 32 | 4
Number analyzed (eyes) | 49 | 6
diopter | -0.75 (0.94) | -0.88 (0.26)

2. Secondary Outcome: Percent of Eyes With Loss of ≥ 2 Lines of Best Spectacle Corrected Visual Acuity (BSCVA)
Time Frame: 6 months
Population: as for baseline characteristics
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Natural Astigmatism | Post Cataract With Residual Astigmatism
Number analyzed (Participants) | 33 | 6
Number analyzed (eyes) | 51 | 10
percentage of eyes | 4.9 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Natural Astigmatism | Post Cataract With Residual Astigmatism
Serious Adverse Events (participants affected / at risk) | 1/34 | 1/6
Other Adverse Events (participants affected / at risk) | 1/34 | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Natural Astigmatism (N=34) | Post Cataract With Residual Astigmatism (N=6)
Hospitalization for auto accident (Surgical and medical procedures) | 1 (1) | 1 (1) — Subject hospitalized after auto accident unrelated to study device or procedure.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Natural Astigmatism (N=34) | Post Cataract With Residual Astigmatism (N=6)
Ocular Penetration (Eye disorders) | 1 (2) | 0 (0)
Possible Allergy to Preservative in Ocular Medication (Immune system disorders) | 0 (0) | 1 (1) — Subject demonstrated possible allergic response to standard postoperative eye drops which was eliminated by changing to a different type of eye drops.

LIMITATIONS AND CAVEATS:
BSCVA determination in eyes with progressing cataracts was sometimes unevaluable, although data are shown as reported.

The number of eyes in "Post Cataract Surgery with Astigmatism" Arm was small, limiting data analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All proposed submissions for publication or presentation of Trial data must be approved by the Sponsor prior to submission. Under no circumstances shall the Investigator(s) publish or disclose data without the Sponsor's written approval.